CLINICAL TRIAL: NCT00004213
Title: An Open Label, Dose Escalation Study to Evaluate Safety, Tolerability, and Pharmacokinetics of 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone (3-AP) in Cancer Patients Using a Single Daily Dose for Five Days
Brief Title: 3-Aminopyridine-2-carboxaldehyde Thiosemicarbazone in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-001-2; CDR0000067390 (Registry Identifier: PDQ (Physician Data Query)); NCI-V99-1579
Record Dates: First submitted 2000-01-28; First posted 2004-05-03 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2007-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of 3-aminopyridine-2-carboxaldehyde thiosemicarbazone in treating patients who have solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effects of 3-aminopyridine-2-carboxaldehyde thiosemicarbazone (3-AP) in patients with solid tumors by evaluating the safety and tolerability, maximum tolerated dose (MTD) and recommended dose for Phase II studies, pharmacokinetics, and tumor response.

OUTLINE: This is a dose escalation study. Patients receive 3-aminopyridine-2-carboxaldehyde thiosemicarbazone (3-AP) IV over 2 hours on days 1-5. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 1-6 patients receive escalating doses of 3-AP until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed for 4 weeks or until recovered.

PROJECTED ACCRUAL: Approximately 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant solid tumor that has failed 1 or more conventional treatments or is unlikely to respond to currently available therapies No active CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: WBC greater than 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 2.0 mg/dL AST and ALT no greater than 3 times upper limit of normal (ULN) Alkaline phosphate no greater than 3 times ULN (no greater than 5 times ULN if liver metastases present) Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No myocardial infarction within the past 3 months No symptomatic coronary artery disease or heart block No uncontrolled congestive heart failure Pulmonary: No moderate or severe pulmonary dysfunction Other: Not pregnant or nursing Negative pregnancy test Fertile women must use effective contraception Body weight greater than 50 kg No active infection No mental deficits and/or psychiatric disorders that would preclude study No other life-threatening illness No bleeding disorder (except occult blood from gastrointestinal cancer)

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior growth factor treatment allowed if blood counts normal Chemotherapy: At least 3 weeks since prior chemotherapy and recovered At least 6 weeks since prior nitrosoureas or mitomycin and recovered Prior hydroxyurea allowed and recovered Endocrine therapy: At least 2 weeks since prior hormonal therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No prior radiotherapy to greater than 30% of the bone marrow Surgery: At least 2 weeks since any prior major surgery Other: At least 4 weeks since other prior investigational agents and recovered No other concurrent investigational agents without consent of sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (2):
- United States (2):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Yale Comprehensive Cancer Center, New Haven, Connecticut